CLINICAL TRIAL: NCT00178841
Title: Open Label Pilot Study of Combination Therapy With Rosiglitazone and Bexarotene to Investigate a Possible Synergism in the Treatment of Cutaneous T-Cell Lymphoma
Brief Title: Combination Drug Study of Bexarotene and Rosiglitazone to Treat CTCL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, John Zic, Associate Professor of Medicine/Dermatology, Vanderbilt University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 050416
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Results first posted 2016-02-17 (Estimated); Last update posted 2016-02-17 (Estimated); Status verified 2016-01

CONDITIONS: Cutaneous T-cell Lymphoma; Mycosis Fungoides; Sezary Syndrome
Keywords: Cutaneous T-cell Lymphoma; CTCL; Mycosis Fungoides; Sezary Syndrome; Bexarotene; Targretin; Rosiglitazone; Avandia
MeSH Terms: conditions — Lymphoma, T-Cell, Cutaneous; Mycosis Fungoides; Sezary Syndrome | interventions — Rosiglitazone; Bexarotene

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Rosiglitazone and Bexarotene — rosiglitazone added to bexarotene capsules

SUMMARY:
The purpose of this trial is to determine if combination therapy with rosiglitazone and bexarotene might have a synergistic effect in the treatment of patients with CTCL.

DETAILED DESCRIPTION:
Treatment options for CTCL include both skin-directed and systemic therapies. Topical treatments are effective for early-stage disease that is localized to the skin. However, disease involving the lymph nodes or visceral sites can be palliated but rarely cured, even with the most aggressive regimens of systemic chemotherapy. Unfortunately, current treatment options at this stage only provide a short term response. Thus, it is important that additional therapies are investigated to manage this malignancy.

Bexarotene has been approved by the FDA for the treatment of Cutaneous T-Cell Lymphoma (CTCL).Bexarotene binds the RXR(Retinoid X Receptor)inside the cell, a receptor that forms heterodimers with a multitude of other nuclear receptors. One of these is the PPARγ (Peroxisome Proliferator Activator Receptor Gamma), a nuclear receptor that binds Rosiglitazone.Rosiglitazone is an FDA approved antidiabetic agent of the Thiazolidinedione class. Rosiglitazone increases insulin sensitivity and is useful in the treatment of type 2 diabetes. In vitro data suggest that rosiglitazone and bexarotene may act synergistically to induce apoptosis in cell lines derived from patients with cutaneous T cell lymphoma (CTCL). This pilot study will investigate this possible synergism in a small cohort of patients with stable or progressive CTCL already being treated with bexarotene.

ELIGIBILITY:
Inclusion Criteria:

* Patients with biopsy proven persistent or recurrent cutaneous cell lymphoma (CTCL) Stage IA-IVA
* Patients with a pathologic proven diagnosis of CTCL that is documented in the patient history.
* Patient has preserved organ function.
* Patient has an ECOG performance status between 0 - 2.
* Women of childbearing potential should be screened for pregnancy prior to treatment and utilize effective contraceptive methods (e.g. barrier) during treatment period.
* Patients over the age of 18 who are willing and able to provide Informed Consent
* The patient has been taking Targretin capsules for at least the last 4 months and the dose has remained relatively stable.
* The patient has had stable or progressive disease over the past 4 months.
* Patient has adequate laboratory parameters for liver and kidney function.

Exclusion Criteria:

* Patients with CD30+ Anaplastic Large Cell Lymphoma
* Patients with pathology consistent with peripheral T-cell lymphoma.
* Patients with Stage IVB (visceral involvement with CTCL).
* Patients with history of Human Immunodeficiency Virus (HIV), Hepatitis B or Hepatitis C infection.
* Patients with a diagnosis of congestive heart failure.
* Patients exhibiting significant edema or unstable cardiovascular disease.
* Patients with a fasting triglyceride level greater then 500mg/dl.
* Patients that have started any new treatment for CTCL in the past 4 months.
* Pregnant women will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2005-06; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John A Zic, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

REFERENCES:
- [Background] Bunn PA Jr, Hoffman SJ, Norris D, Golitz LE, Aeling JL. Systemic therapy of cutaneous T-cell lymphomas (mycosis fungoides and the Sezary syndrome). Ann Intern Med. 1994 Oct 15;121(8):592-602. doi: 10.7326/0003-4819-121-8-199410150-00007. PMID 8085692
- [Background] Koh HK, Charif M, Weinstock MA. Epidemiology and clinical manifestations of cutaneous T-cell lymphoma. Hematol Oncol Clin North Am. 1995 Oct;9(5):943-60. PMID 8522490
- [Background] Duvic M, Hymes K, Heald P, Breneman D, Martin AG, Myskowski P, Crowley C, Yocum RC; Bexarotene Worldwide Study Group. Bexarotene is effective and safe for treatment of refractory advanced-stage cutaneous T-cell lymphoma: multinational phase II-III trial results. J Clin Oncol. 2001 May 1;19(9):2456-71. doi: 10.1200/JCO.2001.19.9.2456. PMID 11331325
- [Background] Zhang C, Ni X, Konopleva M, Andreeff M, Duvic M. The novel synthetic oleanane triterpenoid CDDO (2-cyano-3, 12-dioxoolean-1, 9-dien-28-oic acid) induces apoptosis in Mycosis fungoides/Sezary syndrome cells. J Invest Dermatol. 2004 Aug;123(2):380-7. doi: 10.1111/j.0022-202X.2004.23207.x. PMID 15245439
- [Background] Carr A, Workman C, Carey D, Rogers G, Martin A, Baker D, Wand H, Law M, Samaras K, Emery S, Cooper DA; Rosey investigators. No effect of rosiglitazone for treatment of HIV-1 lipoatrophy: randomised, double-blind, placebo-controlled trial. Lancet. 2004 Feb 7;363(9407):429-38. doi: 10.1016/S0140-6736(04)15489-5. PMID 14962523
- [Background] Wang TD, Chen WJ, Lin JW, Chen MF, Lee YT. Effects of rosiglitazone on endothelial function, C-reactive protein, and components of the metabolic syndrome in nondiabetic patients with the metabolic syndrome. Am J Cardiol. 2004 Feb 1;93(3):362-5. doi: 10.1016/j.amjcard.2003.10.022. PMID 14759393
- [Background] Raji A, Seely EW, Bekins SA, Williams GH, Simonson DC. Rosiglitazone improves insulin sensitivity and lowers blood pressure in hypertensive patients. Diabetes Care. 2003 Jan;26(1):172-8. doi: 10.2337/diacare.26.1.172. PMID 12502676
- [Background] Demierre MF, Tien A, Miller D. Health-related quality-of-life assessment in patients with cutaneous T-cell lymphoma. Arch Dermatol. 2005 Mar;141(3):325-30. doi: 10.1001/archderm.141.3.325. PMID 15781673
- [Background] Bunn PA Jr, Lamberg SI. Report of the Committee on Staging and Classification of Cutaneous T-Cell Lymphomas. Cancer Treat Rep. 1979 Apr;63(4):725-8. No abstract available. PMID 445521
- [Background] Willemze R, Kerl H, Sterry W, Berti E, Cerroni L, Chimenti S, Diaz-Perez JL, Geerts ML, Goos M, Knobler R, Ralfkiaer E, Santucci M, Smith N, Wechsler J, van Vloten WA, Meijer CJ. EORTC classification for primary cutaneous lymphomas: a proposal from the Cutaneous Lymphoma Study Group of the European Organization for Research and Treatment of Cancer. Blood. 1997 Jul 1;90(1):354-71. PMID 9207472
- [Background] Shapiro PE. Advances in the histologic diagnosis of cutaneous T-cell lymphoma. Adv Dermatol. 1996;11:255-84; discussion 285. No abstract available. PMID 8718481
- See also: Pubmed link to article — http://www.ncbi.nlm.nih.gov/pubmed/17184879

RESULTS

PARTICIPANT FLOW:
Groups:
- Rosiglitazone and Bexarotene: Patients maintained their dose of bexarotene during the study and added rosiglitazone. The initial dose of rosiglitazone was 4 mg once daily. If patients showed no response after 1 month and experienced no adverse effects, the dose was increased to a maximum of 8 mg once daily. Dose reductions of rosiglitazone or bexarotene were allowed during the study, but only if necessary to control AEs.
Period: Overall Study
Arm/Group | Rosiglitazone and Bexarotene
Started | 4
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Single Arm Study: All enrolled patients received rosiglitazone in addition to oral bexarotene
Arm/Group | Single Arm Study
Number analyzed (Participants) | 4
Age, Continuous [Median (Full Range); unit: years] | 53 [50 to 66]
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a 50% Improvement in Baseline Skin Score
Description: mSWAT scoring. Range 0 to 400. Measured every 4 weeks.
Time Frame: 16 weeks
Measure: Number; unit: participants
Groups:
- Rosiglitazone and Bexarotene: All 4 enrolled patients received rosiglitazone in addition to oral bexarotene.
Arm/Group | Rosiglitazone and Bexarotene
Number analyzed (Participants) | 4
participants | 0

2. Secondary Outcome: Quality of Life Evaluations
Description: FACT-G, Functional Assessment of Cancer Therapy-General (quality-of-life scale) 0= worst 108=best
Time Frame: baseline and every 4 weeks
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Rosiglitazone and Bexarotene
Number analyzed (Participants) | 4
units on a scale | 86.25 [0 to 108]

3. Secondary Outcome: Pruritus Score
Description: 10-cm visual analog scale, 10= worst, 1=best
Time Frame: 16 weeks
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Rosiglitazone and Bexarotene
Number analyzed (Participants) | 4
units on a scale | 5.7 [0 to 10]

ADVERSE EVENTS:
Time Frame: 2 years
Groups:
- Rosiglitazone and Bexarotene: All enrolled patients received rosiglitazone in addition to oral bexarotene.
Arm/Group | Rosiglitazone and Bexarotene
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 4/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rosiglitazone and Bexarotene (N=4)
Hypertriglyceridemia and hypercholesterolemia (Metabolism and nutrition disorders) | 4 (4) — Hypertriglyceridemia and hypercholesterolemia, two expected adverse events (AEs), were limited to grade 1 because of aggressive management using omega 3 fatty acids, long-acting niacin, fenofibrate, ezetimibe, and statins (N=4).
Anemia (Blood and lymphatic system disorders) | 2 (2)
Neutropenia (Blood and lymphatic system disorders) | 3 (3) — N=2 grade 3 neutropenia
Lymphopenia (Blood and lymphatic system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No